CLINICAL TRIAL: NCT05104164
Title: Prospective and Multicenter Study to Assess the Safety and Effectiveness of a Physiotherapy Treatment Through Self-myofascial Release With Foam Roller in Patients With Hemophilic Ankle Arthropathy. A Randomized Clinical Trial.
Brief Title: Self-myofascial Release in Hemophilic Ankle Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: He-FoamAnk
Record Dates: First submitted 2021-10-25; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia
Keywords: Hemophilic arthropathy; Ankle; Self-myofascial release; Safety; Joint pain; Functionality
MeSH Terms: conditions — Hemophilia A; Arthralgia

STUDY DESIGN:
Masking Description: The physiotherapist in charge of the evaluations was blinded to the conditions and study objectives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-myofascial release (Experimental): Each session will last approximately 15 minutes, with five physiotherapy sessions taking place over a period of 3 months. The Self-Myofascial release protocol for the lower limbs using a Foam Roller and and Solid Ball Massage, adapted to patients with hemophilic ankle arthropathy will include 11 exercises that must be administered bilaterally. A mobile application will be developed where each patient will be able to observe the exercises to be carried out.
  Interventions: Other: Self-myofascial release

INTERVENTIONS:
Other: Self-myofascial release — At home, the patients performed a daily session, lasting 15 minutes each, over 8 weeks. Patients accessed an ad hoc mobile application designed by the Hemophilia Physiotherapy research group (He-Foam®). This app, accessible from any smartphone, made it possible to watch the videos with all the exercises included in the intervention. The seven exercises under the specific protocol for patients with hemophilic arthropathy were: Self-release of the plantar region of the foot with a foam ball; Release of the posterior region of the leg with the foam roller; Release of the anterior leg region with a foam roller; Release of the hamstrings region with a foam roller; Release of adductor muscles with a foam ball; Release of abductor muscles with a foam roller; Release of pelvic trochanteric muscles with a foam roller

SUMMARY:
Introduction: Hemophilic ankle arthropathy is manifested by degenerative functional alterations (deficit of muscle strength, mobility and proprioception) (intra-articular alterations) and chronic pain. Myofascial release techniques are used to treat soft tissue adhesions, relieve pain and reduce tissue sensitivity.

Design. A randomized clinical trial. Aimed: To evaluate the safety and effectiveness of a protocol by self-myofascial release with Foam Roller applied in patients with hemophilic ankle arthropathy.

Patients: 70 patients with ankle arthropathy will be recruited for inclusion in the study. Patients will be recruited in 5 centers, from different regions of Spain.

Intervention: Each session will last approximately 15 minutes, with five physiotherapy sessions per week for a period of 3 months. Patients will be evaluated at baseline, after the intervention, and after a follow-up period of 3 months. The treatment program includes 11 exercises that must be administered bilaterally. A mobile application will be developed where each patient will be able to observe the exercises to be carried out.

Measuring instruments and study variables: digital goniometer (ankle range of motion); visual analog scale and pressure algometer (joint pain); Haemophilia Joint Health Score (joint status); dynamometer assess (muscle strength); 6-Minute Walking test (functionality of lower limbs); Mobile device (Activity record); Finger-floor test (muscle flexibility). At the same time, the study will allow to determine joint bleeding caused by applied physiotherapy treatment.

Expected results: To demonstrate the safety of this Physiotherapy technique in patients with hemophilia. Likewise, an improvement in ankle pain, functionality and joint motion is expected.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Patients with a medical diagnosis of hemophilia A or B.
* Patients with a severe phenotype of hemophilia (<1% FVIII/FIX).
* Patients with a medical diagnosis of hemophilic ankle arthropathy and more than 3 points on the Hemophilia Joint Health Score.
* Nno scheduled orthopedic surgeries during the study phase.
* Signing the informed consent document.

Exclusion Criteria:

* Patients with ankle hemarthrosis in the month before the beginning of the study.
* Patients unable to walk even with technical aids.
* Patients with hemophilic elbow arthropathy that prevented the performance of the exercises.

  * Patients failing to complete at least 80% of the sessions scheduled in the intervention

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline ankle bleeding after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  The safety of the intervention was evaluated through periodic monitoring of the development of ankle hemarthrosis. The physiotherapist in charge of evaluating the patients performed weekly follow-up telephone calls during the experimental phase to evaluate the development of ankle hemarthrosis or other complications (bruising). Bleeding-related data were collected by the evaluator after the follow-up period.

SECONDARY OUTCOMES:
Change from baseline ankle pain after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  The intensity of joint pain was assessed using the visual analog scale (VAS). This scale rates ankle joint pain with scores from zero to 10 points (from no pain to the maximum perceived pain).
Change from baseline range of ankle motion after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  The range of ankle motion in dorsal and plantar flexion was measured with a universal goniometer, with one-degree increments. The patient was placed in a supine position, with the axis of the goniometer on the lateral malleolus and the fixed arm of the goniometer parallel to the fibula. This procedure was accompanied by verbal stimulus to the patient to control the compensatory movement of the toes and the range of movement of the talocrural joint. The unit of measurement is the degrees (the higher the mark, the better the range of motion).
Change from baseline functional capacity after treatment and at 3 months | Screening visit, within the first seven days after treatment and after three months follow-up visit
  Functional capacity was measured with the 6-Minute Walk test, using the standardization described by the American Thoracic Society. The test was performed on a flat, hard, straight, 20-m long surface. Before the test, the evaluator instructed each patient to walk the track twice to familiarize themselves with the test and warm up. The evaluating physiotherapist used standardized verbal stimuli during the test with all subjects. Patients were asked to walk at a constant speed, without jumping or running, for 6 minutes. To measure the exact distance walked during the test the physiotherapist closely followed the patients with a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No